CLINICAL TRIAL: NCT02394652
Title: The Potential for Metformin to Improve Tumor Oxygenation in Locally Advanced Cervix Cancer: A Phase II Randomized Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CXMET1
Record Dates: First submitted 2015-03-16; First posted 2015-03-20 (Estimated); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Uterine Cervical Neoplasms; Squamous Cell Carcinoma; Adenocarcinoma; Carcinoma, Adenosquamous
MeSH Terms: conditions — Uterine Cervical Neoplasms; Carcinoma, Squamous Cell; Adenocarcinoma; Carcinoma, Adenosquamous | interventions — Metformin; Cisplatin; fluoroazomycin arabinoside

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Metformin with Standard Chemoradiation (Experimental): Metformin: About 1 week prior to the start of chemoradiation, take 850 mg of metformin, orally, once a day for 3 days, followed by 850 mg twice a day and continued for the duration of external radiation.
  Chemoradiation: Cisplatin will be given intravenously at 40 mg/m2 week for 5 doses, concomitantly with external beam radiation.
  FAZA-PET scan at baseline and after about 1 week of metformin (just prior to the start of chemoradiation)
  Interventions: Drug: Metformin; Drug: Cisplatin; Drug: FAZA
- Standard Chemoradiation (Active Comparator): Chemoradiation: Cisplatin will be given intravenously at 40 mg/m2 week for 5 doses, concomitantly with external beam radiation.
  FAZA-PET scan at baseline and about 1 week later (just prior to the start of chemoradiation).
  Interventions: Drug: Cisplatin; Drug: FAZA

INTERVENTIONS:
Drug: Metformin — Metformin is an antidiabetic agent given orally.
  Arms: Experimental: Metformin with Standard Chemoradiation
Drug: Cisplatin — Cisplatin is an antineoplastic agent given intravenously.
Drug: FAZA — FAZA is an investigational imaging agent for positron emission tomography scans indicated for hypoxia.
  Other Names: 18F-Fluoroazomycin arabinoside

SUMMARY:
Cervical cancer remains an important health problem worldwide. Poor tumor oxygenation (hypoxia) is associated with inferior survival in cervical cancer and resistance to radiation treatment. Hypoxia-modifying therapies improve survival, but existing therapies are impractical and/or toxic. Metformin, a non-toxic drug for diabetes, has been shown to decrease tumor hypoxia in animal studies and its use is associated with better survival in diabetic cancer patients. It is hypothesized that metformin may decrease cervical tumor hypoxia and thereby improve tumor response to radiation and survival in patients with locally advanced cervix cancer.

This is a randomized, multicenter phase II study of standard chemoradiation in combination with metformin versus standard chemoradiation alone in women with locally advanced cervix cancer. Women randomized to the metformin group will take metformin starting 1 week prior to standard chemoradiation and throughout the duration of external radiation treatment. Tumor hypoxia will be measured by a special X-ray test called positron emission test (PET) performed with a hypoxia dye called FAZA. The main purpose of this study is to see if metformin decreases tumor hypoxia measured on FAZA-PET; information about response and side effects will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed squamous cell carcinoma, adenocarcinoma or adenosquamous carcinoma of the cervix, FIGO stage IB2-IVA
* Planned for radical radiotherapy and concurrent cisplatin chemotherapy.
* Able to receive weekly cisplatin.
* No prior anticancer treatment for cervical cancer
* ECOG 0 or 1
* Life expectancy of greater than 3 months.
* Normal organ and marrow function
* Able to take oral medications.
* Ability to understand and willing to sign the consent form
* Willing to undergo biopsies of cervical tumor.

Exclusion Criteria:

* Evidence of distant metastases
* Receiving any other investigational agents concurrently or within 4 weeks.
* Known diabetes mellitus.
* Currently taking metformin, sulfonylureas, thiazolidinediones or insulin.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to metformin or cisplatin.
* Any condition associated with increased risk of metformin-associated lactic acidosis
* Uncontrolled inter-current illness
* Pregnant women
* History of another invasive malignancy, except for non-melanoma skin cancer or tumors curatively treated with no evidence of disease for >=5 years.
* Known HIV-positive
* History of bowel obstruction or malabsorption syndromes
* History of active clinically significant bleeding
* Contraindications to radiotherapy
* Taking drug disulfiram (antabuse).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-05-21 (Actual); Primary Completion 2021-01-12 (Actual); Study Completion 2021-01-12 (Actual)

PRIMARY OUTCOMES:
• Change in fractional hypoxic volume of the tumor on FAZA-PET scan before and after 1 week of metformin. | About 7 days

SECONDARY OUTCOMES:
Disease-free survival | 2 years
Acute and late gastrointestinal and genitourinary toxicities following metformin and chemoradiation. | 2 years
Effect of metformin on endogenous hypoxia and other markers. | About 7 days
Biomarkers of response to metformin. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Han, M.D., Principal Investigator — Princess Margaret Cancer Centre
Locations (5):
- Canada (5):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Hôpital Maisonneuve-Rosemont, Montreal, Quebec
  - Centre Hospitalier De L'Université de Montréal, Montreal, Quebec